CLINICAL TRIAL: NCT06150586
Title: The PALISA Study - Pain Assessment During Less-Invasive-Surfactant-Administration
Brief Title: Pain Assessment During Less-Invasive-Surfactant-Administration
Acronym: PALISA
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: PALISA
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Infant, Premature, Diseases; Respiratory Distress Syndrome; Surfactant Deficiency Syndrome Neonatal; Pain; Stress
Keywords: Less-Invasive-Surfactant-Administration; Skin Conductance; Neonatal Pain and Sedation Scale; Analgosedation; General stress-level
MeSH Terms: conditions — Infant, Premature, Diseases; Respiratory Distress Syndrome; Pulmonary Atelectasis; Pain | interventions — Weights and Measures; Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants with minimal gestational age of 27 weeks requiring LISA: LISA will be preformed according to our local standard protocol while measuring skin conductance via a specific monitor. At the same time a video is recorded for later unblinded and blinded N-PASS assessment.
  Interventions: Other: Skin Conductance (SC) Measurement; Other: Video Recording

INTERVENTIONS:
Other: Skin Conductance (SC) Measurement — SC will be measured using a specific monitor and three self-adhesive electrodes on one foot of the infant (one plantar and two on the ankles). Peaks per second (the rate of firing in the sympathetic nerves), average amplitude (mean peaks) and area under curve (forcefulness of sympathetic nerve firing) will be automatically analyzed. Corresponding data will be transferred to a separate tablet computer via bluetooth.
Other: Video Recording — The video recording for later N-PASS assessment will be done by a camera fixed above the incubator / resuscitation unit, not interfering with the LISA procedure. The video will show the full body of the newborn as well as the hands / forearms of the treating clinical team with the awareness and oral consent of the treating team.

SUMMARY:
Primary aims of the study are to evaluate the feasibility of Skin conductance (SC) measurements and its correlation to Neonatal Pain and Distress Scale (N-PASS) - scores during the Less-Invasive-Surfactant-Administration (LISA)-procedure in preterm infants. Secondary aims are to evaluate the effect of LISA on the general stress-level in preterm infants with respiratory distress syndrome.

The assessment of pain and stress with SC measurement in addition to the subjective assessment with N-PASS may provide more conclusive data on the sensation of pain or stress during the LISA procedure and therefore the necessity of analgosedation. Therefore, this study might help to identify those infants in need for analgosedation, which would allow an individualized approach in the future.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≥27 0/7 weeks of gestation at birth
* Need for surfactant therapy via LISA according to the local standard operating procedure
* ≥27 0/7 weeks of gestation,
* within first 48 hours of life
* FiO2 ≥0.30 to maintain SpO2 ≥90% for 15 min,
* non-invasive respiratory support with PEEP 6-8 cmH2O
* consent of attending NICU staff for videorecording

Exclusion Criteria:

* Primary intubation in the delivery room
* Severe congenital malformation or other conditions requiring immediate endotracheal intubation
* Insufficient language skills (German or English) of the parents to understand and consent the participation in the study.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infants with ≥27 0/7 weeks of gestation at birth who meet the inclusion criteria and who do not fulfill the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Median peaks per second at prespecified time-points adjusted for median peaks per second at baseline | 2 minutes before LISA, during LISA, 1 hour (±10 minutes) after LISA
  The prespecified time-points are:
  1. baseline: before starting of interventions (2 minutes recording without any intervention);
  2. insertion of nasopharyngeal tube;
  3. insertion of laryngoscope for visualization of the vocal cords;
  4. insertion of LISA catheter
  5. administration of surfactant
  6. removal of catheter
  7. 5 minutes after removal of catheter (2 minutes recording without any intervention)
  8. 1 hour (±10 minutes) after LISA (2 minutes recording without any intervention)

SECONDARY OUTCOMES:
Median Neonatal Pain, Agitation and Sedation Scale (N-PASS) at prespecified time-points, adjusted for median N-PASS at baseline | 2 minutes before LISA, during LISA, 1 hour (±10 minutes) after LISA
  The N-PASS serves as a tool for evaluating pain and sedation levels in newborns. In the context of this study, the focus is solely on assessing pain. Five criteria, including crying, behavior, facial expression, extremity tone and vital signs, are rated on a scale of 0 to 2 points each. These individual scores are then added up to calculate a total pain score, which falls within the range of 0 to 10. A higher total score correlates with a higher level of perceived pain.
  The prespecified time-points, at which the N-PASS will be assessed, are:
  1. baseline: before starting of interventions
  2. during insertion of laryngoscope for visualization of the vocal cords
  3. administration of surfactant
  4. 5 minutes after removal of catheter
  5. 1 hour (±10 minutes) after LISA
Absolute number of apneas | During LISA procedure
  Absolute number of apneas requiring non-invasive pressure ventilation or increase of peak inspiratory pressure or frequency during the LISA procedure
Absolute number of desaturations | During LISA procedure
  Absolute number of decreasing SpO2 requiring increase of FiO2 during the LISA procedure
Absolute number of bradycardia | During LISA procedure
  Absolute number of bradycardia (<100/min) during the LISA procedure
Absolute number of arterial hypotension | During LISA procedure
  Absolute number of arterial hypotension with mean blood pressure lower than gestational age during the LISA procedure
Absolute number of blunt surfactant reflux | During LISA procedure
  Absolute number of blunt surfactant reflux seen in mouth or nose without laryngoscopy during the LISA procedure
Difference in maximum peaks per second before and after apnea | During LISA procedure
  Difference in maximum peaks per second before and after apnea requiring non-invasive pressure ventilation or increase of peak inspiratory pressure or frequency during the LISA procedure
Difference in median peaks per second during 20-second interval before and after apnea | During LISA procedure
  Difference in median peaks per second during 20-second interval before and after apnea requiring non-invasive pressure ventilation or increase of peak inspiratory pressure or frequency during the LISA procedure
Difference in maximum peaks per second before and after desaturation | During LISA procedure
  Difference in maximum peaks per second before and after decreasing SpO2 requiring increase of FiO2 during the LISA procedure
Difference in median peaks per second during 20-second interval before and after desaturation | During LISA procedure
  Difference in median peaks per second during 20-second interval before and after decreasing SpO2 requiring increase of FiO2 during the LISA procedure
Difference in maximum peaks per second before and after bradycardia | During LISA procedure
  Difference in maximum peaks per second before and after bradycardia (<100/min) during the LISA procedure
Difference in median peaks per second during 20-second interval before and after bradycardia | During LISA procedure
  Difference in median peaks per second during 20-second interval before and after bradycardia (<100/min) during the LISA procedure
Difference in maximum peaks per second before and after arterial hypotension | During LISA procedure
  Difference in maximum peaks per second before and after arterial hypotension with mean blood pressure lower than gestational age during the LISA procedure
Difference in median peaks per second during 20-second interval before and after arterial hypotension | During LISA procedure
  Difference in median peaks per second during 20-second interval before and after arterial hypotension with mean blood pressure lower than gestational age during the LISA procedure
Difference in maximum peaks per second before and after blunt surfactant reflux | During LISA procedure
  Difference in maximum peaks per second before and after blunt surfactant reflux seen in mouth or nose without laryngoscopy during the LISA procedure
Difference in median peaks per second during 20-second interval before and after blunt surfactant reflux | During LISA procedure
  Difference in median peaks per second during 20-second interval before and after blunt surfactant reflux seen in mouth or nose without laryngoscopy during the LISA procedure
Difference in heart-rate between baseline and prespecified time-points as listed above. | 2 minutes before LISA, during LISA, 1 hour (±10 minutes) after LISA
  Difference in heart-rate between baseline and prespecified time-points as listed above 2 minutes before LISA, during LISA and 1 hour (±10 minutes) after LISA
Difference in oxygen saturation between baseline and prespecified time-points as listed above. | 2 minutes before LISA, during LISA, 1 hour (±10 minutes) after LISA
  Difference in oxygen saturation between baseline and prespecified time-points as listed above 2 minutes before LISA, during LISA and 1 hour (±10 minutes) after LISA
Difference in SpO2/FiO2-ratio between baseline and prespecified time-points as listed above. | 2 minutes before LISA, during LISA, 1 hour (±10 minutes) after LISA
  Difference in SpO2/FiO2-ratio between baseline and prespecified time-points as listed above 2 minutes before LISA, during LISA and 1 hour (±10 minutes) after LISA
Difference of SpO2/FiO2-ratio compared to skin conductance peaks per second | 2 minutes before LISA, 5 minutes after removal of catheter, 60 Minutes after LISA
  Difference of SpO2/FiO2-ratio at baseline, 5 minutes after removal of catheter and 60 minutes after LISA compared to skin conductance peaks per second (median peaks per second of 2 minute intervals).
LISA failure | Within 24 hours after LISA
  Incidence of LISA failure defined as intubation or repeated LISA within 24 hours
Intubation <72 hours after the LISA procedure | Within 72 hours after LISA
  Incidence of intubation within <72 hours after the LISA procedure
Air-leaks <72 hours after the LISA procedure | Within 72 hours after LISA
  Incidence of air-leaks within <72 hours after the LISA procedure
Incidence of intraventricular hemorrhage | 72 hours after LISA
  Incidence of intraventricular hemorrhage at first ultrasound scan after 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bassler, MD, Study Chair — Newborn Research, Department of Neonatology, University Hospital and University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson J, den Boer MC, Roehr CC. To Sedate or Not to Sedate for Less Invasive Surfactant Administration: An Ethical Approach. Neonatology. 2021;118(6):639-646. doi: 10.1159/000519283. Epub 2021 Oct 8. PMID 34628413
- [Background] Tribolet S, Hennuy N, Snyers D, Lefebvre C, Rigo V. Analgosedation before Less-Invasive Surfactant Administration: A Systematic Review. Neonatology. 2022;119(2):137-150. doi: 10.1159/000521553. Epub 2022 Feb 4. PMID 35124678
- [Background] Hummel P, Puchalski M, Creech SD, Weiss MG. Clinical reliability and validity of the N-PASS: neonatal pain, agitation and sedation scale with prolonged pain. J Perinatol. 2008 Jan;28(1):55-60. doi: 10.1038/sj.jp.7211861. Epub 2007 Oct 25. PMID 18165830
- [Background] Hummel P, Lawlor-Klean P, Weiss MG. Validity and reliability of the N-PASS assessment tool with acute pain. J Perinatol. 2010 Jul;30(7):474-8. doi: 10.1038/jp.2009.185. Epub 2009 Nov 19. PMID 19924132
- [Background] Munsters J, Wallstrom L, Agren J, Norsted T, Sindelar R. Skin conductance measurements as pain assessment in newborn infants born at 22-27 weeks gestational age at different postnatal age. Early Hum Dev. 2012 Jan;88(1):21-6. doi: 10.1016/j.earlhumdev.2011.06.010. Epub 2011 Jul 20. PMID 21764228
- [Background] Storm H. Skin conductance and the stress response from heel stick in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 Sep;83(2):F143-7. doi: 10.1136/fn.83.2.f143. PMID 10952711
- [Background] Storm H. Changes in skin conductance as a tool to monitor nociceptive stimulation and pain. Curr Opin Anaesthesiol. 2008 Dec;21(6):796-804. doi: 10.1097/ACO.0b013e3283183fe4. PMID 18997532
- [Background] Morgan ME, Kukora S, Nemshak M, Shuman CJ. Neonatal Pain, Agitation, and Sedation Scale's use, reliability, and validity: a systematic review. J Perinatol. 2020 Dec;40(12):1753-1763. doi: 10.1038/s41372-020-00840-7. Epub 2020 Oct 2. PMID 33009491
- [Result] Dirler C, Boos V, Bassler D, Benke-Bruderer S, Held U, Ruegger CM, Muehlbacher T. Pain Assessment During Less Invasive Surfactant Administration Using Skin Conductance: A Prospective Cohort Study. Pediatr Res. 2025 Dec 22. doi: 10.1038/s41390-025-04703-9. Online ahead of print. PMID 41429954